CLINICAL TRIAL: NCT07214818
Title: Efficacy of Sodium-Glucose Cotransporter 2 Inhibitors in Adult Patients With Nephrotic Syndrome: A Randomized Controlled Trial
Brief Title: SGLT2 Inhibitors in Adult Primary Nephrotic Syndrome
Acronym: SGLT2-NS
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Maged Saleh Mohsen Ban Hariz, Pharmacist, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MS.25.08.3285
Record Dates: First submitted 2025-10-06; First posted 2025-10-09 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Nephrotic Syndrome
Keywords: SGLT2 inhibitors; Dapagliflozin; Empagliflozin; Proteinuria; Primary Nephrotic Syndrome
MeSH Terms: conditions — Nephrotic Syndrome; Proteinuria | interventions — dapagliflozin; empagliflozin; Standard of Care

STUDY DESIGN:
Intervention Model Description: This interventional study will use a parallel assignment model with three treatment arms:
  Dapagliflozin plus standard therapy. Empagliflozin plus standard therapy. Standard therapy alone (control).
  Randomization will be employed to allocate participants to one of the three groups in a 1:1:1 ratio. Due to the nature of the interventions, this is an open-label study, and blinding will not be feasible.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Dapagliflozin + Standard of Care (Experimental)
  Interventions: Drug: Dapagliflozin; Other: Standard Therapy
- Empagliflozin + Standard of Care (Experimental)
  Interventions: Drug: Empagliflozin; Other: Standard Therapy
- Standard of Care Only (Active Comparator): Standard treatment protocol(institutional standared) for 6 months without any additional SGLT2 inhibitor.
  Interventions: Other: Standard Therapy

INTERVENTIONS:
Drug: Dapagliflozin — Dapagliflozin 10 mg PO once daily for 6 months
  Arms: Dapagliflozin + Standard of Care
Drug: Empagliflozin — Empagliflozin 10 mg PO once daily for 6 month
  Arms: Empagliflozin + Standard of Care
Other: Standard Therapy — immunosuppressive therapy and renoprotective agents for 6 months

SUMMARY:
This randomized controlled clinical trial aims to evaluate the efficacy and safety of sodium-glucose cotransporter 2 (SGLT2) inhibitors (dapagliflozin and empagliflozin) in adult patients with primary nephrotic syndrome. The study will compare three groups: dapagliflozin plus standard therapy, empagliflozin plus standard therapy, and standard therapy alone.

The primary objective is to assess whether SGLT2 inhibitors reduce proteinuria, maintain remission, and prevent relapse. Secondary objectives include evaluating effects on kidney function (eGFR, serum creatinine) and monitoring safety outcomes.

Participants will continue their baseline standard care and will be followed for 6 months with regular clinical evaluations, laboratory tests, and adverse event monitoring.

DETAILED DESCRIPTION:
This randomized, controlled, open-label, single-center clinical trial is designed to investigate the efficacy and safety of sodium-glucose cotransporter 2 (SGLT2) inhibitors, specifically dapagliflozin and empagliflozin, in adult patients with primary nephrotic syndrome (PNS).

Primary nephrotic syndrome is characterized by significant proteinuria, hypoalbuminemia, and related complications. While traditional therapies such as corticosteroids and immunosuppressive agents remain the cornerstone of treatment, their limited efficacy and adverse effects highlight the need for novel therapeutic options. Evidence from large clinical trials has shown that SGLT2 inhibitors improve renal outcomes in patients with chronic kidney disease and type 2 diabetes; however, their role in primary nephrotic syndrome patients has not been fully established.

In this trial, eligible participants will be adults (≥18 years) with biopsy-confirmed primary nephrotic syndrome and an estimated glomerular filtration rate (eGFR) ≥25 mL/min/1.73m². Patients with secondary causes of nephrotic syndrome (e.g., diabetic nephropathy, lupus nephritis, amyloidosis), significant liver impairment, or contraindications to SGLT2 inhibitors will be excluded.

Participants will be randomized into three groups:

Group A: Dapagliflozin 10 mg once daily plus standard therapy. Group B: Empagliflozin 10 mg once daily plus standard therapy. Group C: Standard therapy alone (control).

All groups will continue to receive stable doses of background immunosuppressive therapy and renoprotective agents as part of standard of care.

The study duration will be 6 months. Baseline demographics, clinical data, and laboratory parameters will be collected. Follow-up assessments will include proteinuria (urine protein-to-creatinine ratio), serum albumin, serum creatinine, eGFR, uric acid, total cholestrol, liver enzyme(AST,ALT), TNF-α, complete blood count and serum sugar level. Clinical outcomes such as remission, relapse, and adverse events will be recorded.

The primary outcomes are changes in proteinuria, TNF-α levels, and rates of remission and relapse. Secondary outcomes include changes in kidney function (serum creatinine, eGFR), safety profile, and treatment compliance.

This study is expected to provide novel insights into the therapeutic role of SGLT2 inhibitors in primary nephrotic syndrome and may guide future clinical practice in the management of this condition.

ELIGIBILITY:
Inclusion Criteria:

Adult patients (≥18 years). Biopsy-confirmed primary nephrotic syndrome (e.g., idiopathic membranous nephropathy, minimal change disease, focal segmental glomerulosclerosis).

Estimated glomerular filtration rate (eGFR) ≥25 mL/min/1.73m² using CKD-EPI formula.

On stable dose of immunosuppressive therapy and renoprotective agents for ≥4 weeks prior to randomization.

Able to signed informed consent.

Exclusion Criteria:

Diagnosis of secondary nephrotic syndrome as : diabetes mellitus, lupus nephritis, and amyloidosis.

* Impaired liver functions (ALT or AST values exceeding 3 folds upper limit of normal (ULN) at the screening visit).
* Glomerular hematuria (red blood cells more than ten cells per high power field (HPF) after routine urinalysis for more than three times in the last 2 weeks).
* History of severe hypersensitivity or contraindications to dapagliflozin or empagliflozine.
* Pregnancy or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-11-15 (Actual); Primary Completion 2026-07-05 (Estimated); Study Completion 2026-09-06 (Estimated)

PRIMARY OUTCOMES:
1. Change in Proteinuria (uPCR) | Baseline to 6 months
  Change from baseline in urine protein/creatinine ratio
Change in TNF-α Levels | Baseline to 6 months
  Change in serum TNF-α measured by ELISA as an exploratory biomarker.

SECONDARY OUTCOMES:
Change in Estimated Glomerular Filtration Rate (eGFR) | Baseline to 6 months
  Mean change in eGFR calculated by CKD-EPI formula.
Incidence of Adverse Events | Throughout the 6-month study perio
  Frequency and severity of adverse effects including infection, gastrointestinal upset, oral candidiasis, and other safety concerns.
Treatment Compliance | Up to 6 months
  Proportion of participants with documented adherence to study medication and standard therapy.
Remission Rate | Up to 6 months
  Proportion of patients achieving remission
Relapse Rate | Up to 6 months
  Proportion of patients experiencing relapse

CONTACTS AND LOCATIONS:
Overall Officials: Moetaza M Soliman, Associate Professor, Study Chair — Clinical Pharmacy and Pharmacy Practice Department, Faculty of Pharmacy, Mansoura University; Mustafa O Sharaf El-Deen, Lecturer, Study Director — Clinical Pharmacy and Pharmacy Practice Department, Faculty of Pharmacy, Mansoura University
Locations (1):
- Urology & Nephrology Center, Mansoura University, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No